CLINICAL TRIAL: NCT02514655
Title: Role of a Simple Mechanical Device of Pressure Control in the Balloon of the Endotracheal Tube to Prevent Ventilator-acquired Pneumonia
Brief Title: Simple Mechanical Device to Control Pressure in the Balloon of the Endotracheal Tube to Prevent Ventilator-acquired Pneumonia
Acronym: PAV-PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P111113; 2014-A00190-47 (Other: Eudract CT)
Record Dates: First submitted 2015-07-07; First posted 2015-08-04 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2023-08

CONDITIONS: Mechanical Ventilation; Tracheal Intubation; Ventilator-acquired Pneumonia; Intubation -Related Tracheal Lesions
Keywords: Tracheal intubation; Cuff pressure; Ventilator-acquired pneumonia; Intensive care unit; Tracheal injuries
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Nosten® monitoring (Experimental): One experimental group with the control of the cuff pressure by Nosten® device
  Interventions: Device: Nosten® pressure control (it's not an antibiotic, but simple device)
- 2: Manual monitoring (Active Comparator): One control group with the manual monitoring of the cuff pressure and inflation of the balloon
  Interventions: Other: Manual pressure control

INTERVENTIONS:
Device: Nosten® pressure control (it's not an antibiotic, but simple device) — One experimental group with the control of the cuff pressure by Nosten® device
  Arms: 1: Nosten® monitoring
Other: Manual pressure control — One control group with the manual monitoring of the cuff pressure and inflation of the balloon
  Arms: 2: Manual monitoring

SUMMARY:
Hypothesis: Nosten® device is able to reduce the time of underinflated balloon and removes excess pressure. This device may thus reduce the risk of ventilator-acquired pneumonia (VAP) and early tracheal lesions resulting from intubation with decreased discomfort, morbidity, and nursing workload.

The main objective of the investigators is to show that Nosten® device is more effective than monitoring and manual inflation of the balloon of the tracheal tube to prevent VAP occurrence.

DETAILED DESCRIPTION:
Multicenter, controlled, prospective randomized open study with blinded assessment of the primary endpoint. Two groups are set up: one experimental group with the control of the cuff pressure by the Nosten® device versus one control group with the manual monitoring of the cuff pressure and inflation of the balloon.

Inclusion: All orotracheally intubated patients for an expected period > 48 hours will be selected. Inclusion will be decided using an algorithm adapted to each center to limit the number of inclusion per month without any biases.

The total number of required insclusion is 500, or 250 / group. This calculation is based on the assumption that a frequency of 25% of patients having at least one VAP in the reference strategy, ensuring a 80% power in the detection by Chi-2 test with a difference 10%. A bilateral risk of first species determined at 5% was considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients admitted in the ICU, mechanically ventilated and whose trachea was intubated by the oral route using tubes with catheter polyvinyl chloride "high-volume low pressure" and of standard shape tubes Intubation indication is decided by the physicians in charge according to the usual criteria of respiratory, neurological and /or hemodynamic failure
* With an expected duration of mechanical ventilation > 48 hours

Exclusion Criteria:

* Patients intubated by nasotracheal route
* Patients with tracheotomy before admission
* Patients intubated with a polyurethane balloon catheter or a polyvinyl chloride balloon catheter of conical shape
* Previously intubated patients for > 48 hours before their possible recruitment
* Moribund patients (terminal illness or care-limiting decision)
* Minors protected or incapacitated patients
* Patients with recently diagnosed ENT cancer
* Patients with facial, thoracic, spinal or upper airway trauma
* Patients burned, intoxicated by fire fumes or caustic ingestion
* Patient pregnant or breastfeeding (or with known positive urine pregnancy test before inclusion)
* Patient intubated with a subglottic suction tube
* Unaffiliated patients to a social security
* Patients included in any other scientific study that may interfere with the outcome criteria of this study. This includes any other study on tracheal intubation or mechanical ventilation, if the use of the pressure control device may interfere with its endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-08-15 (Actual); Primary Completion 2015-08-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of the incidence of VAP as defined according to the criteria of the American Thoracic Society (3 months after inclusion) | up to 3 months
  To prove that the Nosten® device is more effective than monitoring and manual inflation of the catheter balloon in reducing the occurrence of VAP.

SECONDARY OUTCOMES:
Reduction in the tracheobronchial bacterial colonization assessed using the bacteriological examination of the tracheal aspiration (as long as the patient is intubated during 3 months after inclusion) | up to 3 months
  using the bacteriological examination of the tracheal aspiration during the intensive care hospitalization
Reduction of clinically suspected Ventilator-Acquired Pneumonia (VAP) | up to 3 months
  before obtaining microbiological results needed to affirm the Ventilator-Acquired Pneumonia (VAP) according to the criteria of the American Thoracic Society (3 months)
Reduction in the duration of antibiotic therapy administered to patients, if diagnosed with ventilator-aquired-pneumonia (VAP) (3 months) | up to 3 months
  Reduction of clinically suspected Ventilator-Acquired Pneumonia (VAP)
Reduction in the periods of hyper-pressure and under-inflation (as long as the patient is intubated during 3 months after inclusion) | up to 3 months
  Using Nosten® device
Reduction in the significant early laryngeal and tracheal injuries related to intubation (3 months) | up to 3 months
  using the tracheal ischemia score [Touat L. Intensive Care Med 2014]

CONTACTS AND LOCATIONS:
Overall Officials: Bruno MEGARBANE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Réanimation Médical et Toxicologique, Paris, France